CLINICAL TRIAL: NCT02616094
Title: Multimodal Neuroimaging of Stress and Reward Cues to Assess Alcoholism Risk and Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1501015225; 2R01AA013892-11 (NIH)
Record Dates: First submitted 2015-11-16; First posted 2015-11-26 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Seeking Alcohol Dependent Adults (Experimental): Group consists of 100 treatment seeking alcohol dependent (AD) men and women (ages 18-60). AD subjects will complete either 8 weeks of outpatient treatment at the Yale Stress Center, or the first 4 weeks as inpatient treatment at the CNRU, followed by 4 weeks of outpatient treatment at the Yale Stress Center. While in outpatient treatment, AD subjects may be admitted to the CNRU or HRU for the 1-5 days prior to one or both of their scans, to ensure abstinence for their scans.
  Interventions: Device: Multi-method Neuroendocrine and Neuroimaging Procedure Scan 1; Device: Multi-method Neuroendocrine and Neuroimaging Procedure Scan 2
- Social Drinking Controls (Active Comparator): Group consists of demographically and handedness matched 50 socially drinking controls. Healthy controls will be moderate and binge/heavy social drinkers who will participate in a single MRI session after baseline assessments. Healthy controls may be admitted to the HRU overnight prior to their scan.
  Interventions: Device: Multi-method Neuroendocrine and Neuroimaging Procedure Scan 1
- Prazosin/Placebo Group (Active Comparator): This is a separate group of 60 treatment seeking AD subjects in a NIAAA-funded RCT of Prazosin vs placebo for alcohol dependence ( PI: Sinha, Hic protocol 0705002691, NCT00585780) to assess target primary and secondary predictors of alcohol treatment outcomes in the context of a currently ongoing RCT. AD subjects enrolled in the PZ/PL RCT will NOT be given drugs as part of this study. That study and intervention is listed elsewhere (NCT00585780). Subjects will participate in a baseline scan and a second scan between weeks 10-12 of the 12-week RCT with follow-ups. PZ/PL is only given to subjects enrolled in 0705002691, not the current protocol.
  Interventions: Device: Multi-method Neuroendocrine and Neuroimaging Procedure Scan 1; Device: Multi-method Neuroendocrine and Neuroimaging Procedure Scan 2

INTERVENTIONS:
Device: Multi-method Neuroendocrine and Neuroimaging Procedure Scan 1 — The MRI scan will be conducted on a 3-T Siemens Trio MRI system equipped with a standard quadrature head coil, using T1 MPRAGE sequence for structural scanning and T2*-sensitive gradient-recalled single shot echo planar pulse sequence for functional scans. Two multimethod MRI scans will be conducted in the AD sample, while the controls will participate in a single scan.
Device: Multi-method Neuroendocrine and Neuroimaging Procedure Scan 2 — The MRI scan will be conducted on a 3-T Siemens Trio MRI system equipped with a standard quadrature head coil, using T1 MPRAGE sequence for structural scanning and T2*-sensitive gradient-recalled single shot echo planar pulse sequence for functional scans. Two multimethod MRI scans will be conducted in the AD sample, while the controls will participate in a single scan.
  Arms: Prazosin/Placebo Group; Treatment Seeking Alcohol Dependent Adults

SUMMARY:
Extending previous findings, and applying a novel multi-method translational approach, this project hypothesizes that there are alcohol-related neuroendocrine and neural changes observable in acute and protracted abstinence, and which can accurately classify future relapse and treatment outcome in separate alcohol dependent (AD) patient samples, thereby validating them as biomarkers of relapse, with potential clinical utility as prognostic markers in identifying and treating those most susceptible to relapse.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, aged 18-60 years;
* Good health as verified by screening examination;
* Able to read English and complete study evaluations;
* Able to provide informed written and verbal consent;
* AD sample must meet DSM-5 criteria for AUD as assessed using SCID-I and have positive alcohol urine toxicology screens on admission to study; while HC group must never have met criteria for AUD, with non-binging and nonhazardous alcohol intake levels( men: below15 drinks/week; women: less than 8 drinks/week); and with negative alcohol urine toxicology screens; Page

Exclusion Criteria:

* Meet current criteria for dependence on another psychoactive substance, excluding nicotine; (ii) Current use of opiates or past history of opiate abuse/dependence;
* Regular use of anticonvulsants, sedatives/hypnotics, prescription analgesics, other antihypertensives, anti-arrhythmics, antiretroviral medications, SSRI's naltrexone, antabuse;
* Psychotic or otherwise severely psychiatrically disabled (i.e., suicidal, homicidal, current mania);
* Significant underlying medical conditions such as a history of seizure disorder, cerebral, renal, thyroid or cardiac pathology which in the opinion of study physician would preclude subjects from fully cooperating or be of potential harm during the course of the study;
* Any psychotic disorder or current Axis I psychiatric symptoms (excluding anxiety disorders) requiring specific attention, including need for psychiatric medications;
* hypotensive individuals with sitting blood pressure below 90/50 mmHG;
* Women who are pregnant, nursing or refuse to use a reliable form of birth control (as assessed by pregnancy tests during initial medical evaluation, and assessed every two weeks during the course of the study); and
* those with metal in their body excluded from MRI due to safety.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Time to Relapse | Up to 200 days
  The Time-Line Follow-Back Interview will be used to assess alcohol use in the previous ninety days, during the study and during follow-up until relapse occurs or 200 days is up.

SECONDARY OUTCOMES:
Time to heavy drinking relapse | Up to 200 days
  The Time-Line Follow-Back Interview will be used to assess alcohol use in the previous ninety days (this is standard for TLFB surveys), during the study and during follow-up until relapse occurs or 200 days is up.
Percent of days of alcohol use in follow-up | Up to 200 days
  The Time-Line Follow-Back Interview will be used to assess alcohol use in the previous ninety days (which is standard for TLFB surveys), during the study and during follow-up. This can only be measured once relapse occurs. It will be measured once relapse occurs or will not be measured at all if relapse does not occur within 200 days.

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Stress Center, New Haven, Connecticut, United States